CLINICAL TRIAL: NCT06001268
Title: Support Through Remote Observation and Nutrition Guidance Program for Individuals With Pancreatic Cancer Undergoing Surgery (STRONG-PCS)
Brief Title: Support Through Remote Observation and Nutrition Guidance Program (STRONG-PCS)
Acronym: STRONG-PCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22476
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer
Keywords: Nutrition Support
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRONG-PCS Intervention (Experimental): Participants will receive an initial in-person consultation with a dietician within 2 weeks of hospital discharge. Then participants will receive individually tailored, bi-weekly nutrition counseling from a dietician via telehealth or in person and remote monitoring through a smart phone app and wearable sensor to allow participants to log food intake while sharing their data with a dietician.
  Interventions: Behavioral: Fitbit Data Collection; Behavioral: Nutrition Counseling; Behavioral: Survey
- Usual Care (Active Comparator): Participants will be referred for nutrition counseling from a dietitian based on clinical discretion.
  Interventions: Behavioral: Nutrition Counseling; Behavioral: Survey

INTERVENTIONS:
Behavioral: Fitbit Data Collection — Participants will log food intake while sharing their data with a dietician in real time for 12 weeks
  Arms: STRONG-PCS Intervention
Behavioral: Nutrition Counseling — Participants will receive individually tailored, bi-weekly nutrition counseling from a dietician via telehealth or in person.
Behavioral: Survey — Participants will take a survey at baseline and weeks 4,8,& 12. (FACT-G) Questionnaire includes questions about participant's physical, social, emotional and functional well being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher total score indicates better quality of life.

SUMMARY:
The purpose of the study is to assess the feasibility and participant satisfaction with the Support through Remote Observation and Nutrition Guidance program. The program provides enhanced dietician access and nutrition support for participants living with pancreatic cancer who are undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Diagnosis of pancreatic cancer
* Completed open pancreatic surgery (e.g., Whipple, distal/subtotal pancreatectomy, total pancreatectomy) for treatment at Moffitt Cancer Center
* Discharged on an oral diet
* Able to speak and read English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* Determined to be ineligible for surgery during evaluation (e.g., cancer metastasis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate - Feasibility | Up to 48 months
  The study will be deemed feasible if ≥ 50% of eligible participants are enrolled.
Retention Rate - Feasibility | at 8 weeks
  The study will be deemed feasible if ≥ 70% of participants enrolled at baseline will be retained at 8 weeks.
Data Collection - Feasibility | at 8 weeks
  The study will be deemed feasible if ≥ 70% of participants log food for greater than 80% of study days.
Participant Satisfaction - Acceptability | at 8 weeks
  The study will be deemed acceptable if ≥ 70% of participants rate the overall intervention as satisfactory using a validated 4-item scale (score range 0-20, score >/= 12).
Participant Rating on Ease of Use the Mobile Application - Usability | at 8 weeks
  The study will be deemed usable if ≥ 60% of participants rate the mobile application as easy-to-use for logging dietary intake using a validated 10-item scale (score range from 0-100, score of >/=60).

SECONDARY OUTCOMES:
Malnutrition-Significant weight loss | 90 days
  Significant weight loss is defined as >5% and >10% of body weight at 30, 60, and 90 days after discharge. This will be calculated based on weight obtained during clinic visits.
Malnutrition - Low BMI | at Baseline, 30, 60 and 90 days
  Low BMI will be defined as <20kg/m² for individuals <70 years old and <22kg/m2 for individuals ≥70 years old. This will be calculated based on weight and height measurements from clinic visits.
Malnutrition - Low Skeletal Muscle Mass | At baseline, 30, 60 and 90 days
  Low muscle mass will be estimated by calculating skeletal muscle index (SMI) from routinely collected CT scans at baseline and 90 days after discharge (CT scans are conducted every 3 months). Low muscle mass will be defined as SMI ≤38.9 cm2 /m2 for females and SMI ≤55.4 cm2 /m2 for males.
Quality of Life | at Baseline, 4, 8 and 12 weeks
  Quality of Life will be measured using the Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire includes questions about the participant's physical, social, emotional and functional well being over the past 7 days. This questionnaire uses a 5 point Likert-type scale, 0=not at all, 4=very much. A higher score indicates a better quality of life.
Hospital Readmissions | 30, 60 and 90 days post-hospital discharge
  Hospital readmissions will be measured using a self-reported survey item to determine whether the patient was admitted to the index hospital or another hospital after hospital discharge.
Malnutrition -Nutritional Status | at Baseline, 30, 60 and 90 days
  Nutritional status will be measured using the Patient-Generated Subjective Global Assessment (PG-SGA) Short Form (score range: 0-35) and categorized based on a prior validation study (0-1 well nourished, 2-8 at-risk, = 9 severely malnourished).

CONTACTS AND LOCATIONS:
Overall Officials: Kea Turner, PhD, Principal Investigator — Moffitt Cancer Center; Pamela J Hodul, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner K, Milano J, Santiago C, Coutinho J, Sprow O, Hume E, Nardella N, Alishahi Tabriz A, Islam JY, Hodul PJ. A patient-mediated strategy to improve nutrition care after transition from hospital to home for pancreatic cancer surgery: a pilot randomised controlled trial study protocol. BMJ Open. 2026 Jan 28;16(1):e113207. doi: 10.1136/bmjopen-2025-113207. PMID 41605580